CLINICAL TRIAL: NCT07203885
Title: Prospective Studies on Artificial Intelligence for Cancer Pathology Evaluation
Brief Title: AI-Assisted Acute Myeloid Leukemia Evaluation With the Leukemia End-to-End Analysis Platform (LEAP) Versus Clinician-Only Assessment
Acronym: LEAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard Medical School (HMS and HSDM) (Other)
Collaborators: National Taiwan University Hospital (Other); Far Eastern Memorial Hospital (Other); Taipei Veterans General Hospital, Taiwan (Other Government); Brigham and Women's Hospital (Other); Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Kun-Hsing Yu, Associate Professor of Biomedical Informatics, Harvard Medical School (HMS and HSDM)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Diagnostic
Other Study IDs: IRB23-0403
Record Dates: First submitted 2025-09-08; First posted 2025-10-02 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Acute Promyelocytic Leukemia (APL); Acute Myeloid Leukaemia (AML)
Keywords: AI-Assisted Detection; Acute Promyelocytic Leukemia; Bone Marrow Slide; Whole-slide images; Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Promyelocytic, Acute; Leukemia, Myeloid, Acute

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Unaided Review First, Then AI-Assisted Review (Active Comparator): Readers first complete Block X (Unaided) on their assigned subset SX (34 slides). They then complete Block Y (AI-Assisted) on two separate subsets: SY1 (34 slides; AI as Double-Check) and SY2 (34 slides; AI as First Look). Within Block Y, the order of Y1 and Y2 is randomized. For each reader, SX, SY1, and SY2 are disjoint and stratified by APL status.
  Interventions: Behavioral: Unaided Review First, Then AI-Assisted Review
- AI-Assisted Review First, Then Unaided Review (Active Comparator): Readers first complete Block Y (AI-Assisted) on two assigned subsets: SY1 (34 slides; AI as Double-Check) and SY2 (34 slides; AI as First Look), with the order of Y1 and Y2 randomized. They then complete Block X (Unaided) on subset SX (34 slides). For each reader, SX, SY1, and SY2 are disjoint and stratified by APL status.
  Interventions: Behavioral: AI-Assisted Review First, Then Unaided Review

INTERVENTIONS:
Behavioral: Unaided Review First, Then AI-Assisted Review — Readers first complete Block X (Unaided) on their assigned subset SX (34 slides). They then complete Block Y (AI-Assisted) on two separate subsets: SY1 (34 slides; AI as Double-Check) and SY2 (34 slides; AI as First Look). Within Block Y, the order of Y1 and Y2 is randomized. For each reader, SX, SY1, and SY2 are disjoint and stratified by APL status.
  Arms: Unaided Review First, Then AI-Assisted Review
Behavioral: AI-Assisted Review First, Then Unaided Review — Readers first complete Block Y (AI-Assisted) on two assigned subsets: SY1 (up to 40 slides; AI as Double-Check) and SY2 (up to 40 slides; AI as First Look), with the order of Y1 and Y2 randomized. They then complete Block X (Unaided) on subset SX (up to 40 slides). For each reader, SX, SY1, and SY2 are disjoint and stratified by APL status.
  Arms: AI-Assisted Review First, Then Unaided Review

SUMMARY:
This study will test whether artificial intelligence (AI) can help doctors diagnose a rare blood cancer called acute promyelocytic leukemia (APL) more quickly and accurately. Doctors usually examine bone marrow samples under a microscope to make this diagnosis, but it can be challenging and time-consuming.

In this study, doctors will review bone marrow samples under three different conditions:

* Unaided Review: Without AI assistance.
* AI as Double-Check: AI-generated evaluation shown after the doctor makes an initial decision.
* AI as First Look: AI-generated evaluation shown at the start of the review.

Doctors will be randomly assigned to different orders of these three conditions. This design will allow us to compare how AI support affects diagnostic accuracy, speed, and confidence.

DETAILED DESCRIPTION:
This study aims to evaluate the effect of artificial intelligence (AI) assistance on clinicians' diagnostic performance in detecting acute promyelocytic leukemia (APL) using Wright-Giemsa-stained bone marrow whole-slide images (WSIs). The Leukemia End-to-End Analysis Platform (LEAP) will serve as the AI model under assessment.

This is a single-session, within-reader study. Participants will be randomly assigned to one of two study arms, which differ in the order of diagnostic blocks:

* Arm 1 (X -> Y): Block X (Unaided Review): Clinicians review WSIs without AI support. Diagnostic accuracy, time to decision, and confidence will be recorded.

Block Y (AI-Assisted Review): Comprising two sub-blocks presented in randomized order:

Y1 (AI as Double-Check): Clinicians provide an initial diagnosis and confidence score without the aid of AI. AI predictions are then revealed, and clinicians may revise their diagnosis. Both pre-AI and post-AI decisions will be recorded.

Y2 (AI as First Look): Clinicians review WSIs with AI-predicted diagnoses visible from the beginning.

* Arm 2 (Y -> X): Block Y (AI-Assisted Review): Sub-blocks Y1 and Y2 presented in randomized order.

Block X (Unaided Review): As described above.

Each clinician will review 102 de-identified WSIs. For each reader, slides will be randomly divided into three disjoint subsets (e.g. 34/34/34), stratified by APL status, and assigned to Block X (Unaided), Block Y1 (AI as Double-Check), or Block Y2 (AI as First Look). No slide will be shown to the same reader in more than one block.

In addition, the AI system will independently generate diagnostic predictions for all WSIs to enable benchmarking; however, this does not constitute a participant arm.

Ground-truth diagnoses will be determined by molecular confirmation and expert consensus.

ELIGIBILITY:
Inclusion Criteria for Pathology Slides (i.e., Cases):

* Wright-Giemsa-stained bone marrow aspirate smears
* Final diagnosis confirmed through molecular testing in conjunction with expert pathology evaluation

Exclusion Criteria for Pathology Slides (i.e., Cases):

* Poor-quality or unreadable slides
* Cases used in AI training

Inclusion Criteria for Readers (i.e., Participants):

* Board-certified or board-eligible pathologists, or board-certified/board-eligible hematologists who routinely make hematopathology diagnoses in their clinical practice
* Willingness to complete both unaided and AI-assisted review sessions

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2025-09-09 (Actual); Primary Completion 2025-10-10 (Actual); Study Completion 2025-10-10 (Actual)

PRIMARY OUTCOMES:
Diagnostic performance of APL detection | Periprocedural (at the time of slide review)
  Performance of clinicians (unaided and AI-assisted) in detecting APL, measured in accuracy, sensitivity, specificity, positive predictive value, and negative predictive value.

SECONDARY OUTCOMES:
Time to diagnosis | Periprocedural (at the time of slide review)
  Average time (seconds per case) required to finalize a diagnosis.
Inter-observer variability | Periprocedural (at the time of slide review)
  Agreement among clinicians across conditions, measured using inter-rater reliability metrics (e.g., kappa statistics).
Concordance between AI predictions and clinicians' diagnoses | Periprocedural (at the time of slide review)
  The proportion of cases in which AI predictions match clinicians' decisions in each study condition.
Decision-change rates | Periprocedural (at the time of slide review)
  The proportion of cases in which a clinician's initial diagnosis is revised after exposure to AI assistance.
Net benefit after AI exposure | Periprocedural (at the time of slide review)
  The overall change in diagnostic accuracy attributable to AI assistance.
Clinician confidence level | Periprocedural (at the time of slide review)
  Self-reported diagnostic confidence recorded for each case.
  Scale:
  5 - Absolutely Certain; 4 - Mostly Certain; 3 - Unsure; 2 - Very Doubtful;
  1 - Random Guess;
  With 5 being the highest confidence score and 1 being the lowest.

CONTACTS AND LOCATIONS:
Locations (1):
- Harvard Medical School, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-10-29): https://cdn.clinicaltrials.gov/large-docs/85/NCT07203885/Prot_SAP_000.pdf